CLINICAL TRIAL: NCT07186400
Title: Beyond Straight Lines: The Test-retest Reliability and Concurrent Validity of the Figure of Eight Walk Test and the 360° Turn Test in Patients With Total Hip Arthroplasty
Brief Title: The Test-retest Reliability and Concurrent Validity of the Figure of Eight Walk Test and the 360° Turn Test
Status: Recruiting | Type: Observational
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Other Study IDs: Test-retest reliability
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Arthroplasty
Keywords: total hip arthroplasty; test-retest reliability; validity; balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Total Hip Arthroplasty: Participants who have undergone total hip arthroplasty and are enrolled to evaluate the reliability and validity of performance-based outcome measures.

SUMMARY:
To the best of the authors' knowledge, there are no existing studies that have evaluated the reliability and validity of the Figure-of-Eight Walk Test (F8WT) and the 360° Turn Test (360°TT) specifically in patients with total hip arthroplasty (PwTHA). The objective of this investigation was to assess the test-retest reliability and concurrent validity of the F8WT and 360°TT within this patient population.

DETAILED DESCRIPTION:
This study involves a cross-sectional design with 54 unilateral PwTHA cases. Assessments to be conducted during the first session include the F8WT, 360°TT, Timed Up and Go (TUG), and Harris Hip Score (HHS). Subsequently, the F8WT and 360°TT will be retested one hour after the initial test. The reliability of these tests will be determined using the intraclass correlation coefficient (ICC). Concurrent validity will be assessed using the Pearson correlation coefficient. Additionally, the standard error of measurement (SEM95) and minimum detectable change (MDC95) will be calculated for the F8WT and 360°TT.

ELIGIBILITY:
Inclusion Criteria:

* surgery performed at least 6 months prior;
* unilateral total hip arthroplasty;
* patients who scored at least 24 points on the Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* a history of additional surgery on the lower extremities;
* bilateral THA or revision surgery;
* severe neurological or orthopedic conditions that may influence musculoskeletal mobility or walking;
* body mass index (BMI) of 40 kg/m² or higher;
* lack of consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have undergone total hip arthroplasty and are enrolled to evaluate the reliability and validity of performance-based outcome measures.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Figure of eight walk test (F8WT) | Baseline
  The F8WT was developed to evaluate parameters such as gait speed, balance, and directional turning capabilities. The protocol involves participants walking in a figure-eight pattern around two cones positioned 1.52 meters apart. Timing commences when participants initiate the task from the midpoint of the figure-eight trajectory and concludes upon their return to the starting location. Participants' walking directions and chosen speeds are adjusted according to individual preferences and comfort levels.
Figure of eight walk test (F8WT) | 1 hour after baseline
  The F8WT was developed to evaluate parameters such as gait speed, balance, and directional turning capabilities. The protocol involves participants walking in a figure-eight pattern around two cones positioned 1.52 meters apart. Timing commences when participants initiate the task from the midpoint of the figure-eight trajectory and concludes upon their return to the starting location. Participants' walking directions and chosen speeds are adjusted according to individual preferences and comfort levels.
360° turn test (360°TT) | Baseline
  The 360°TT serves as a performance evaluation tool aimed at assessing dynamic balance capabilities. The protocol requires participants to execute a complete 360° turn in the shortest possible duration. Turn time and the number of steps employed during the maneuver are recorded using a stopwatch. A turn duration exceeding 2.1 seconds is indicative of a heightened risk of balance deterioration and potential functional impairment.
360° turn test (360°TT) | 1 hour after baseline
  The 360°TT serves as a performance evaluation tool aimed at assessing dynamic balance capabilities. The protocol requires participants to execute a complete 360° turn in the shortest possible duration. Turn time and the number of steps employed during the maneuver are recorded using a stopwatch. A turn duration exceeding 2.1 seconds is indicative of a heightened risk of balance deterioration and potential functional impairment.

SECONDARY OUTCOMES:
Timed up and go test (TUG) | Baseline
  Physical performance will be assessed using the TUG test, which is known for its reliability among PwTHA. The procedure involved standing up from a 45 cm chair, walking along a 3-metre path, turning around, and sitting back down on the chair. It will be used to examine concurrent validity against the F8WT and 360° Turn Test.
Harris hip score (HHS) | Baseline
  The HHS is a comprehensive, multidimensional instrument specifically designed to clinically assess patients with total hip arthroplasty (PwTHA). It consists of four distinct domains: pain, function, deformity, and range of motion (ROM). The total possible score is 100 points, with higher scores indicating better functional status. It will be used to examine concurrent validity against the F8WT and 360° Turn Test.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Dr., Principal Investigator — Artvin Coruh University
Locations (1):
- Zeynep Yıldız Kızkın, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahl JS, Nelson MJ, Taylor M, Solomon LB, Arnold JB, Thewlis D. Biomechanical changes and recovery of gait function after total hip arthroplasty for osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2018 Jul;26(7):847-863. doi: 10.1016/j.joca.2018.02.897. Epub 2018 Feb 21. PMID 29474993
- [Background] Yarar HA, Narin S, Erduran M, Gurbanov I. The test-retest reliability and concurrent validity of 360 degrees turn test in patients with knee osteoarthritis. Somatosens Mot Res. 2024 Jun;41(2):90-96. doi: 10.1080/08990220.2023.2178402. Epub 2023 Feb 14. PMID 36786842
- [Background] Barker KL, Batting M, Schlussel M, Newman M. The reliability and validity of the Figure of 8 Walk test in older people with knee replacement: does the setting have an impact? Physiotherapy. 2019 Mar;105(1):76-83. doi: 10.1016/j.physio.2018.07.003. Epub 2018 Jul 25. PMID 30241701
- [Background] Tillman M, Molino J, Zaferiou AM. Frontal plane balance during pre-planned and late-cued 90 degree turns while walking. J Biomech. 2022 Aug;141:111206. doi: 10.1016/j.jbiomech.2022.111206. Epub 2022 Jun 20. PMID 35772242
- [Background] Almajid R, Goel R, Tucker C, Keshner E. Balance confidence and turning behavior as a measure of fall risk. Gait Posture. 2020 Jul;80:1-6. doi: 10.1016/j.gaitpost.2020.05.020. Epub 2020 May 20. PMID 32454377
- [Background] Mokkink LB, Elsman EBM, Terwee CB. COSMIN guideline for systematic reviews of patient-reported outcome measures version 2.0. Qual Life Res. 2024 Nov;33(11):2929-2939. doi: 10.1007/s11136-024-03761-6. Epub 2024 Aug 28. PMID 39198348
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Ozden F, Ozkeskin M, Ar E, Yuceyar N. Gait assessment in shaped pathways: The test-retest reliability and concurrent validity of the figure of eight test and L test in multiple sclerosis patients without mobility aids. Mult Scler Relat Disord. 2022 Sep;65:103998. doi: 10.1016/j.msard.2022.103998. Epub 2022 Jun 25. PMID 35777291
- [Background] Dobson F, Hinman RS, Hall M, Marshall CJ, Sayer T, Anderson C, Newcomb N, Stratford PW, Bennell KL. Reliability and measurement error of the Osteoarthritis Research Society International (OARSI) recommended performance-based tests of physical function in people with hip and knee osteoarthritis. Osteoarthritis Cartilage. 2017 Nov;25(11):1792-1796. doi: 10.1016/j.joca.2017.06.006. Epub 2017 Jun 22. PMID 28647467
- [Background] Ramadanov N, Voss M, Hable R, Hakam HT, Prill R, Salzmann M, Dimitrov D, Becker R. Postoperative Harris Hip Score Versus Harris Hip Score Difference in Hip Replacement: What to Report? Orthop Surg. 2025 Jan;17(1):3-21. doi: 10.1111/os.14272. Epub 2024 Oct 21. PMID 39434235
- [Background] Celik D, Can C, Aslan Y, Ceylan HH, Bilsel K, Ozdincler AR. Translation, cross-cultural adaptation, and validation of the Turkish version of the Harris Hip Score. Hip Int. 2014 Sep-Oct;24(5):473-9. doi: 10.5301/hipint.5000146. Epub 2014 Sep 10. PMID 25264204
- [Background] Pittenger DJ. Internet research: an opportunity to revisit classic ethical problems in behavioral research. Ethics Behav. 2003;13(1):45-60. doi: 10.1207/S15327019EB1301_08. PMID 14552304
- [Background] Gandhi R, Tsvetkov D, Davey JR, Syed KA, Mahomed NN. Relationship between self-reported and performance-based tests in a hip and knee joint replacement population. Clin Rheumatol. 2009 Mar;28(3):253-7. doi: 10.1007/s10067-008-1021-y. Epub 2008 Oct 8. PMID 18853222